CLINICAL TRIAL: NCT07106580
Title: A Monocentric, Prospective, Randomized, Placebo-controlled, Double-blinded Trial Investigating the Safety and Efficacy of Lyophilized Fecal Microbiota Transplantation Capsules in Decolonization of Patients With Intestinal Carriage of Multidrug-resistant Organisms
Brief Title: Safety and Efficacy of Lyophilized Fecal Microbiota Transplantation Via Capsules for Intestinal Multidrug-resistant Bacteria Decolonization
Acronym: FORCE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Rijeka (Other)
Collaborators: Clinical Hospital Center Rijeka (Other)
Responsible Party: Principal Investigator, Igor Rubinić, Prinicpal investigator, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2170-1-42-04-3/1-25-5
Record Dates: First submitted 2025-07-28; First posted 2025-08-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Colonization, Asymptomatic
Keywords: FMT; Fecal microbiota transplantation; Colonization; MDRO; Multidrug-resistant bacteria; Lyophilization
MeSH Terms: conditions — Asymptomatic Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT (Experimental): lyophilized FMT capsules
  Interventions: Other: lyophilized FMT capsules
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Other: Placebo capsules

INTERVENTIONS:
Other: lyophilized FMT capsules — A total of 18 capsules containing 3060 mg of lyophilizate given through 3 days (three capsules twice daily)
  Arms: FMT
Other: Placebo capsules — 18 capsules of identical appearance and weight given in the same way as FMT capsules
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oral capsules containing lyophilized stool from healthy donors (fecal microbiota transplantation or FMT) can safely and effectively decolonize multidrug-resistant organisms (MDROs) from the intestines in adults. The main questions it aims to answer are:

1. Does FMT via oral capsules reduce or eliminate intestinal MDRO colonization?
2. What side effects or adverse events occur after taking FMT capsules?

Researchers will compare FMT capsules to placebo capsules to see if FMT is effective and safe for decolonizing MDROs.

Participants will:

* Take either FMT capsules or placebo capsules by mouth
* Attend 4 follow-up study visits over 6 months (180 days) for microbiological testing and safety monitoring
* Provide stool samples and report any side effects

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) is a growing global health threat, with multidrug-resistant organisms (MDROs) causing substantial morbidity, mortality, and healthcare costs. Among the most concerning MDROs are extended-spectrum beta-lactamase-producing Enterobacterales (ESBL-E), carbapenem-resistant Enterobacterales (CRE), and vancomycin-resistant enterococci (VRE). Colonization of the intestinal tract with these pathogens significantly increases the risk of subsequent invasive infections and facilitates nosocomial transmission, particularly in high-risk populations such as hospitalized or immunocompromised patients.

Current approaches to MDRO decolonization, including selective digestive decontamination and antimicrobial therapy, have shown inconsistent efficacy and carry the risk of further promoting resistance. Therefore, there is an urgent need for novel, non-antibiotic interventions that can effectively reduce intestinal MDRO colonization.

Fecal microbiota transplantation (FMT) has emerged as a promising strategy to restore a healthy gut microbiome and outcompete resistant organisms. While FMT is an established therapy for recurrent Clostridioides difficile infection, its use in MDRO decolonization remains investigational. Most available data come from small cohort studies or case series, with limited evidence from controlled trials.

This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy and safety of FMT using lyophilized stool capsules for the decolonization of intestinal MDROs.

Study Design and Intervention

Participants will be randomly assigned (1:1) to receive either:

* Intervention arm: Oral FMT capsules containing lyophilized fecal microbiota from healthy screened donors
* Control arm: Oral placebo capsules identical in appearance but containing an inert substance Both participants and investigators will be blinded to the allocation. The capsules will be administered under supervision, and the total number of capsules and dosing schedule will be consistent with existing FMT protocols for recurrent C. difficile infection, adapted as needed for study-specific safety and feasibility.

The study will include 48 adult participants (≥18 years) who have laboratory-confirmed intestinal colonization with one or more MDROs (e.g., ESBL-E, CRE, or VRE). Colonization must be confirmed by at least one positive stool or rectal swab culture within a defined timeframe prior to randomization.

Study Procedures and Timeline

Participants will be monitored over a 180-day follow-up period, including four follow-up study visits:

Screening/Baseline/Intervention (visit 1-3): Informed consent, screening, confirmation of MDRO colonization, baseline characteristics, randomization. The intervention can be started on the same day.

Follow-up consists of several visits: Visit 4 (Day 7±1), 5 (Day 30±3), 6 (Day 90±3), and 7 (Day 180±7). At each visit, stool samples or rectal swabs will be collected for MDRO culture and participants will be assessed for adverse events, new infections, antibiotic use or changes in health status.

Primary and Secondary Objectives Primary objective: To evaluate the efficacy of oral FMT capsules in decolonizing intestinal MDROs at 180 days post-treatment, measured by the absence of target MDROs in stool cultures.

Secondary objectives: To assess the persistence of decolonization at follow-up visits. To evaluate the safety and tolerability of FMT capsules, including the incidence and severity of adverse events. To evaluate the rate of early decolonization (day 30).

Safety Monitoring All participants will be monitored for adverse events, including gastrointestinal symptoms, infections, allergic reactions, and other unexpected events. Any serious adverse events (SAEs) will be reported to the relevant ethics committee and regulatory authorities in accordance with local and international guidelines.

Potential Impact This trial addresses a critical unmet need in infectious disease management and antimicrobial stewardship. If successful, oral FMT capsules could become a scalable, non-antibiotic approach to MDRO decolonization, with important implications for preventing infections, limiting MDRO spread, and reducing the use of broad-spectrum antimicrobials in high-risk populations. Furthermore, the capsule-based delivery offers a patient-friendly, less invasive alternative to colonoscopic or enema-based FMT administration, potentially improving acceptability and adherence.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years,
* rectal swab positive for MDRO (including but not limited to: CRE, ESBL-E, VRE) within a week of randomization,
* capable of swallowing oral capsules,
* willing to give informed consent

Exclusion Criteria:

* antibiotic treatment on the day of inclusion,
* pregnant or breastfeeding, women of childbearing potential who are unwilling or unable to use an acceptable method of birth control,
* patients with terminal diseases with expected life expectancy < 6 months,
* unwillingness to ingest the capsules,
* a history of colectomy, present colostomy or ileostomy,
* patients with the diagnosis/treatment of inflammatory or functional bowel disease,
* patients with malignant bowel diseases,
* absolute neutrophil count < 500/mm3,
* selective digestive decolonization with antibiotics within 6 months before randomization,
* severe allergy to capsule components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy (decolonization on visit 7) | Day 180 ± 7 from randomization
  Decolonization on day 180 as determined by microbiological analysis. Rectal swabs or stool samples will be collected during each of the scheduled visits. Stool samples are preferred and are self-collected by participants. If stool sample is unavailable, a rectal swab will be collected. The samples will be promptly delivered to the local microbiology laboratory and processed using standard laboratory procedures.

SECONDARY OUTCOMES:
Early decolonization | Day 30 +/- 3 after randomization
  The proportion of subjects not carrying MDRO at 30 days after randomization as determined by rectal swab or stool sample culture.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From randomization to day 180 +/-7
  At each study visit, participants will be questioned about adverse events they have experienced since the last study visit. Adverse events are any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. In the absence of reported events, participants will specifically be questioned about common symptoms such as abdominal pain, constipation, nausea, flatulence, vomiting, and febrile episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Center Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the publication (e.g., microbiological results, adverse events, decolonization status) will be made available upon reasonable request. Data will be shared with qualified researchers for academic purposes under a data use agreement. Requests should be directed via e-mail.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Data will be shared with qualified researchers for academic purposes under a data use agreement. Requests should be directed via e-mail.